CLINICAL TRIAL: NCT04907591
Title: Effects of Postoperative Prognosis Management Service Using Mobile Applications and Smart Bands for Gastric Cancer Patients
Brief Title: Postoperative Prognosis Management Service Based mHealth for Gastric Cancer Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Samsung Medical Center (Other)
Collaborators: National IT Industry Promotion Agency (Unknown)
Responsible Party: Principal Investigator, JiHye Hwang, Professor, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: NIPA AIoT_Cancer
Record Dates: First submitted 2021-05-20; First posted 2021-06-01 (Actual); Last update posted 2022-10-26 (Actual); Status verified 2022-10

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Wearable Electronic Devices

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mHealth App and wearable device (Experimental): an intervention group (App+IoT device) uses a smart care application tailored to gastric cancer patients created by reflecting the treatment process immediately after surgery and a wearable smart band for 12 months.
  Interventions: Device: mHealth App and wearable device
- Education brochure (No Intervention): Control group is provided general education through the hospital brochure.

INTERVENTIONS:
Device: mHealth App and wearable device — an intervention group (App+IoT device) uses a smart care application tailored to gastric cancer patients created by reflecting the treatment process immediately after surgery and a wearable smart band worn on wrist for 12 months.
  Arms: mHealth App and wearable device

SUMMARY:
Recently, the use of mobile health is increasing for the purpose of managing prognosis such as recurrence, survival and quality of life by using a wearable smart band together with a smartphone application. In the era of the 4th revolution, mobile health for the purpose of comprehensive prognosis for cancer patients is becoming a very good tool. As a result of applying a mobile application for health management (nutrition, health education, exercise, etc.) to 203 gastric cancer or colon cancer patients undergoing chemotherapy in the previous study, gastric cancer patients are most interested in health-related education and information.

As such, it was possible to confirm the clinical significance of short-term and temporary health care through mobile applications and smart bands during the treatment process for gastric cancer patients, but the study was insufficient to generalize the number of subjects. Therefore, until now, the results of a multicenter randomized-control study have not been found after long-term application as a supportive tool from immediately after surgery (before treatment) to during the treatment process.

Therefore, in gastric cancer patients who need prognosis management after surgery, we will investigate the effect of mobile application with smart band which has a modular structure reflecting the treatment method and treatment process after surgery.

This study targets patients who underwent gastric cancer surgery, an intervention group (App+IoT device) uses a smart care application tailored to gastric cancer patients created by reflecting the treatment process immediately after surgery and a wearable smart band for 12 months. Control group was provided general education through the hospital brochure. Evaluation will be conducted 2-3days after surgery (before discharge), and at 1, 3, 6, and 12 months after surgery.

ELIGIBILITY:
Inclusion Criteria:

* AJCC stage I-III who has undergone radical gastric cancer surgery (chemotherapy, radiation therapy is irrelevant)
* Patients aged 19 to 75 years old
* Those who can use prognosis management applications and can perform regular follow-up inspections outpatients
* Patients carrying Android or iOS smartphones
* Patients who voluntarily decide to participate and give written consent after hearing detailed explanations about this study

Exclusion Criteria:

* Those who have difficulty using gastric cancer applications (exercise performance, diet management, etc.) due to severe underlying diseases, neuromusculoskeletal diseases, cognitive, and visual impairments

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 324 (Estimated)
Dates: Start 2021-05-17 (Actual); Primary Completion 2023-05-30 (Estimated); Study Completion 2024-05-30 (Estimated)

PRIMARY OUTCOMES:
Change of body composition (weight, kg) | between baseline (postoperative 2-3days) and postoperative 6 months
  comparison between groups in change of weight between baseline (postoperative 2-3days) and postoperative 6 months

SECONDARY OUTCOMES:
Change of Quality of life (EORTC-QLQ-C30) | between baseline (postoperative 2-3days) and postoperative 6 months
  comparison between groups in change of quality of life between baseline (postoperative 2-3days) and postoperative day 6 months
  This questionnaire contains 30 items regarding general health status, five functional scales (ie, physical, role, cognitive, emotional, and social functioning), three symptom scales (ie, fatigue, pain, and nausea or vomiting), and six single-item scales (ie, dyspnea, appetite loss, constipation, diarrhea, financial difficulties, and insomnia). Each scale includes a different set of items, which are calculated using specific coding procedures. Higher scores for the general health status and the functional scales imply positive results, whereas the symptom and the single-item scales are interpreted inversely.
Pain (Numeric rating scale, NRS) | Enrollment (postoperative 2-3days), postoperative 1month, 3month, 6month, 12month
  According to time frame with between-group and within group, trends will be found. NRS score (11 point scales) ranges from 0 (no pain) to 10 (possible to image maximum pain). Higher score indicates higher pain.
Self-reported symptom and Quality of life (EORTC-QLQ-STO22) | postoperative 1month, 3month, 6month, 12month
  According to time frame with between-group and within group, trends will be found. EORTC QLQ-STO22 is composed of 5 multi-item scales and 4 single-item measures. For the EORTC QLQSTO22, like symptom scales, a high score represents low QoL.
  This questionnaire evaluates the effect of chemotherapy, radiation therapy on symptom and quality of life. Therefore, from postoperative 1 month, it will be evaluated.
Physical activity (IPAQ-SF) | Enrollment (postoperative 2-3days), postoperative 1month, 3month, 6month, 12month
  According to time frame with between-group and within group, trends will be found. There are two forms of output from scoring the IPAQ. Results can be reported in categories (low activity levels, moderate activity levels or high activity levels) or as a continuous variable (MET minutes a week). MET minutes represent the amount of energy expended carrying out physical activity. Higher METs or category level indicates higher physical activity.
Grip strength | Enrollment (postoperative 2-3days), postoperative 1month, 3month, 6month, 12month
  According to time frame with between-group and within group, trends will be found. Using a grip dynamometer, take three measurements on both hands. Higher value (kg) indicates higher grip strength.
  Since this test is judged to have a mild effect of abdominal pain after surgery, it is evaluated from enrollment.
Lower extremity muscle endurance (30seconds chair stands test) | postoperative 1month, 3month, 6month, 12month
  According to time frame with between-group and within group, trends will be found. It measures the number of times you sit and stand up in a chair for 30 seconds. Higher value (number) indicates higher lower extremity muscle endurance.
  It is judged that the 30seconds chair stands test will be difficult due to abdominal pain after surgery, so the evaluation is performed only at the other F/U points excluding the enrollment date.
2 Minute walk test (2MWT, evaluation of cardiopulmonary endurance) | postoperative 1month, 3month, 6month, 12month
  According to time frame with between-group and within group, trends will be found. The 2MWT is a measurement of endurance that assesses walking distance over two minutes.
  It is judged that the 2MWT will be difficult due to abdominal pain after surgery, so the evaluation is performed only at the other F/U points excluding the enrollment date.
Nutrition assessment (Mini-nutrition assessment, MNA) | Enrollment (postoperative 2-3days), postoperative 1month, 3month, 6month, 12month
  According to time frame with between-group and within group, trends will be found. The short form of the MNA (MNA-SF) is a screening tool consisting of six questions on food intake, weight loss, mobility, psychological stress, or acute disease, the presence of dementia or depression, and body mass index (BMI). The maximum score for this part is equal to 14. A score equal to or higher than 12 indicates that the subject under study has an acceptable nutritional status thus excluding malnutrition and/or malnutrition risk, meanwhile, a score ≤ 11 implicates to proceed with the complete version of the MNA (MNA-LF). This version consists of 12 additional items and provides a maximum possible overall assessment of 30 scores: a score of fewer than 17 indicates malnutrition, a score of 17-23.5 indicates a risk for malnutrition and a score higher 23.5 indicates well-nourishment.
Visceral fat (㎠) | Enrollment (postoperative 2-3days), postoperative 6month, 12month
  According to time frame with between-group and within group, trends will be found.
  Visceral fat at navel level measured by Computed Tomography
Muscle mass (lumbar 2,㎠) | Enrollment (postoperative 2-3days), postoperative 6month, 12month
  According to time frame with between-group and within group, trends will be found.
  Muscle mass at lumbar 2 measured by Computed Tomography

CONTACTS AND LOCATIONS:
Overall Officials: JIHYE HWANG, Professor, Principal Investigator — Physical & Rehabilitation Medicine Samsung Medical Center
Locations (1):
- Korea University Anam Hospital, Seoul, Seongbuk-gu, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kim I, Lim JY, Kim JK, Lee JH, Sohn TS, Park S, Kang SH, Lee JY, Hwang JH. Effectiveness of a personalized digital exercise and nutrition-based rehab program for patients with gastric cancer after surgery: Study protocol for a randomized controlled trial. Digit Health. 2023 Jul 17;9:20552076231187602. doi: 10.1177/20552076231187602. eCollection 2023 Jan-Dec. PMID 37485329